CLINICAL TRIAL: NCT04494958
Title: Phase IB Clinical Trial of Palbociclib and Binimetinib in Advanced Triple Negative Breast Cancer With Hyperactivation of ERK and/or CDK4/6
Brief Title: Palbociclib and Binimetinib in Advanced Triple Negative Breast Cancer
Acronym: PALBOBIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion Oncosur (Network)
Collaborators: Pfizer (Industry); Apices Soluciones S.L. (Industry); Pierre Fabre Ibérica, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALBOBIN; 2020-000930-16 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — palbociclib; binimetinib

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, single-arm, open label, phase IB clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib + Binimetinib (Experimental)
  Interventions: Drug: Combination, Palbociclib + Binimetinib

INTERVENTIONS:
Drug: Combination, Palbociclib + Binimetinib — Patients will then start treatment with continuous oral binimetinib 45 mg/BID and palbociclib 100 mg daily, 21 days on / 7 days off, until disease progression. Study treatment will continue until disease progression.
  If treatment tolerance is good, after a full cycle patients will be allowed to escalate palbociclib to 125 mg, according to the study investigators' decision. Alternatively, patients with non tolerable grade 2 events will resume at 30 mg/BID of binimetinib upon recovery, maintaining palbociclib at 100 mg 21-on/7-off. Depending on the side-effects, in case of clear relationship with palbociclib is established, palbociclib -instead of binimetinib - will be reduced to 75 mg daily.

SUMMARY:
This study is an interventional, prospective, multicentric, single-arm, open label, phase Ib clinical trial. This study will be carried out in patients diagnosed of metastatic or locally advanced unresectable triple negative breast cancer with activation of ERK and/or CDK4/6 in which the following will be assesed: the overall response rate, the aggregation of antitumor effect depending on the different kinome profiles and the safety profile to the combination of palbociclib and binimetinib.

ELIGIBILITY:
Inclusion Criteria:

1. Women >18 years-old.
2. Diagnostic of metastatic or locally advanced non-resectable TNBC.
3. Patient that have received at least one and up to two previous lines of therapy for metastatic TNBC and failed to last treatment. Previous treatments can be of any nature (chemotherapy, immunotherapy, antiangiogenics, experimental therapy, etc.).

   Women with known BRCA1/BRCA2 germline mutations must have received a platinum based treatment or treatment with a PARP inhibitor.
4. Patient must have experienced disease progression to the previous treatment line according to the RECIST 1.1 or iRECIST criteria.
5. Availability of tumor tissue for ERK and CDK4/6 testing is mandatory prior to study inclusion, preferably obtained after last treatment or the most recent sample as possible (from metastatic site or first diagnosis according to sample availability). If the patient has not a tumor sample available prior to study inclusion, the patient will not be allowed to participate in the study.
6. Ability to understand and signing of the written patient information/informed consent form (PIS/ICF) for ERK and CDK4/6 testing. ERK and CDK4/6 testing will be performed centrally at CNIO.
7. Ability to understand and signing the written PIS/ICF for study treatment eligibility. Signed informed consent form must be available before any studyspecific procedure for the respective study parts may begin.
8. Positivity for ERK and/or CDK4/6, defined as showing an H-score above the top-quartile according to published definitions [1].
9. ECOG performance status of 0-1.
10. Evaluable disease according to RECIST 1.1 criteria.
11. Life expectancy >24 weeks.
12. Adequate bone marrow, liver and renal function as assessed by laboratory requirements conducted within 7 days before first study drug administration:

    1. Absolute neutrophil count (ANC) ≥ 1.500/mm3 (without granulocyte colony-stimulating factor support within 2 weeks before the first study drug administration)
    2. Hemoglobin ≥ 9 g/dL (without transfusion or erythropoietin within 4 weeks before the first study drug administration)
    3. Platelet count ≥ 100.000/mm3 (without transfusion within 2 weeks before the first study drug administration)
    4. Total bilirubin ≤ 2 X the upper limit of normal (ULN).
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 X ULN (≤ 5 times ULN for patients with liver metastases)
    6. Glomerular filtration rate (GFR) > 50 mL/min/1.73 m2 according to the modification of diet in renal disease (MDRD) abbreviated formula.
13. Patients must have recovered to ≤ Grade 1 in terms of toxicity from prior treatments (excluding neuropathy which can be ≤ Grade 2, and alopecia).
14. Patients must be able to take oral medications.
15. Patients must have adequate cardiac function, defined as:

    1. Left ventricular ejection fraction (LVEF) > 50% as determined by echocardiogram or multigated acquisition scan (MUGA).
    2. QTc < 480 msec.
16. Negative serum pregnancy test in women of childbearing potential (performed within 7 days before the first treatment). Negative results must be available before the first study drug administration. Pregnancy test will not be performed in postmenopausal women.
17. Women of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period since the signature of the informed consent form and until at least 1 month after the last study drug administration. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements. Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception.Zoledronic acid or denosumab started prior to trial registration is allowed, but in case they are required after initiation of trial procedures, adequate justification is required.

Exclusion Criteria:

1. Participants who have had chemotherapy, radiotherapy, or major surgery within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
2. Patients that received during the metastatic disease setting any of the study drugs, palbociclib or binimetinib.
3. Participants receiving any other study agents concurrently with the study drugs. Zoledronic acid or denosumab for bone metastases, started at least 15 days prior to enrollment are allowed.
4. Participants with symptomatic brain metastases that require chronic steroids. Patients with a history of brain metastases are permitted to enroll as long as they have been treated, are off of steroids, and have been stable for a minimum of one month on imaging.
5. Irradiation of single lesions in the last 28 days prior to trial recruitment, if it is the only location of the disease and it has not progressed. Patients with radiated single lesions that has progressed are allowed.
6. Concurrent use of strong CYP3A4 inhibitors/inducers is prohibited due to drug-drug interactions with palbociclib. Moderate CYP3A4 inhibitors/inducers should be used with caution.
7. Uncontrolled intercurrent illness including, but not limited to:

   1. ongoing or active infection requiring systemic treatment
   2. symptomatic congestive heart failure
   3. cardiac arrhythmia
   4. psychiatric illness/social situations that would limit compliance with study requirements
   5. hypertension, defined as systolic blood pressure > 160 mmHg despite medical management
   6. myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting < 6 months prior to screening
8. History of QT syndrome, Brugada syndrome, known history of QTc prolongation, or Torsades de Pointes.
9. History of Gilbert's syndrome.
10. History of neuromuscular disorders that are associated with elevated CK (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
11. Previous or concurrent cancer except:

    1. cervical carcinoma in situ
    2. treated basal-cell carcinoma or squamous cell skin cancer c. any other cancer curatively treated > 3 years before the first study drug administration
12. Malabsorption syndrome or uncontrolled nausea, vomiting, or diarrhea that may interfere with the absorption of oral study medication in the opinion of the investigator.
13. Pregnant women or breast-feeding.
14. Known HIV-positive individuals on combination antiretroviral therapy.
15. Active hepatitis B virus (HBV; chronic or acute; defined as having a known positive hepatitis B surface antigen [HBsAg] test at the time of screening) or hepatitis C infection requiring treatment.

    1. Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible if HBV DNA is negative.
    2. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Any condition that in the opinion of the investigator would interfere with evaluation of study treatment or interpretation of patient safety or study results, or inability to comply with the study and follow-up procedures.
17. Participation in another clinical study with investigational medicinal products within 4 weeks before the first study drug administration.
18. Clinically active infections within 2 weeks before the first study drug administration.
19. Treatment with therapeutic oral or i.v. antibiotics within 2 weeks before the first study drug administration. Patients receiving prophylactic antibiotics (e.g. for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
20. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
21. Current diagnosis of any retinal disorders including retinal detachment, retinal pigment epithelial detachment (RPED), serous retinopathy or retinal vein occlusion or risk factors for RVO (e.g., uncontrolled glaucoma or history of hyperviscosity or hypercoagulability syndrome).
22. Peripheral sensory neuropathy of CTCAE v.5.0 Grade 2 or higher
23. Major surgery, open biopsy or significant traumatic injury within 4 weeks before the first study drug administration (central line surgery is not considered major surgery).
24. Renal failure requiring peritoneal dialysis or hemodialysis.
25. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In this Case, gender is a eligibility criteria because it is a specific cancer in women.
Enrollment: 24 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel Quintela-Fandino, MD, Principal Investigator — Centro Nacional de Investigaciones Oncológicas
Locations (8):
- Spain (8):
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospìtal Universitario de la Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital QuirónSalud Madrid, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palbociclib + Binimetinib
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Palbociclib + Binimetinib
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1
  Latin | 1
  White | 22
Region of Enrollment [Number; unit: participants]
  Spain | 24

OUTCOME MEASURES:

1. Primary Outcome: 3 Months Progression Free Survival. Probability That the Cancer Has Not Progressed at 3 Months Calculated With Kaplan Meier.
Description: Progression free survival (PFS) is defined as the time from the date of start treatment until objective tumor progression or death from any reason. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment. Progression free survival at three months is provided.
Time Frame: 3 months
Population: All patients includeed in the study that received at least one dose of study treatment and have at least one evaluation visit after received the first dose of treatment.
Measure: Number (95% Confidence Interval); unit: perceent probability at 3 months
Arm/Group | Palbociclib + Binimetinib
Number analyzed (Participants) | 19
perceent probability at 3 months | 15.8 [0.0 to 32.2]

2. Secondary Outcome: Progression Free Survival
Description: Time from the date of first dose of study treatment to the date of progression or death (from any cause).
Time Frame: 3 months
Population: All patients included in this study that received at least one dose of study treatment and have at least one evaluation visit after received the first dose of treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Binimetinib
Number analyzed (Participants) | 19
Months | 1.8 [1.6 to 2.1]

3. Secondary Outcome: Overall Response Rate
Description: Percentage of patients that achieve complete response or partial response according to RECIST 1.1 criteria
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Binimetinib
Number analyzed (Participants) | 19
Participants | 0

ADVERSE EVENTS:
Time Frame: All adverse events that occur during the period comprehended from the start of study treatment to 30 days after last dose of the investigational products were recorded, an average of 3 months.
Arm/Group | Palbociclib + Binimetinib
All-Cause Mortality (participants affected / at risk) | 9/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib + Binimetinib (N=24)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib + Binimetinib (N=24)
Anaemia (Blood and lymphatic system disorders) | 9 (13)
Neutropenia (Blood and lymphatic system disorders) | 12 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5)
Blindness (Eye disorders) | 2 (2)
Ocular toxicity (Eye disorders) | 2 (2)
Retinopathy (Eye disorders) | 2 (2)
Scintillating scotoma (Eye disorders) | 3 (6)
Vision blurred (Eye disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 17 (28)
Gingival bleeding (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Stomatitis (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 17 (25)
Chest pain (General disorders) | 3 (3)
Mucosal inflammation (General disorders) | 4 (10)
Oedema (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 7 (10)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (3)
COVID-19 (Infections and infestations) | 3 (4)
Overdose (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Blood creatine phosphokinase increased (Investigations) | 5 (8)
Ejection fraction decreased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 5 (6)
Platelet count decreased (Investigations) | 6 (10)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 10 (22)
Lymphoedema (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04494958/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT04494958/SAP_001.pdf